CLINICAL TRIAL: NCT04907682
Title: Pharmacokinetics, Tolerability and Safety of Favipiravir Compared to Ribavirin for the Treatment of Lassa Fever: A Randomized Controlled Open Label Phase II Clinical Trial
Brief Title: Pharmacokinetics, Tolerability and Safety of Favipiravir Compared to Ribavirin for the Treatment of Lassa Fever
Acronym: SAFARI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bernhard Nocht Institute for Tropical Medicine (Other Government)
Collaborators: University of Hamburg-Eppendorf (Other); Alliance for International Medical Action (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Bordeaux (Other); Federal Medical Centre, Owo (Industry); Irrua Specialist Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAFARI; PACTR202010817169062 (Registry Identifier: Pan African Clinical Trials Registry)
Record Dates: First submitted 2021-05-06; First posted 2021-06-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-11

CONDITIONS: Lassa Fever
Keywords: Ribavirin; Favipiravir; viral hemorrhagic fever
MeSH Terms: conditions — Lassa Fever; Hemorrhagic Fevers, Viral | interventions — favipiravir

STUDY DESIGN:
Intervention Model Description: Exploratory, prospective, controlled, multisite, open label, randomized clinical trial with two arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous ribavirin (Active Comparator): standard treatment: Irrua regimen
  * 100 mg/kg Day 1 (dose is divided: 2/3 stat, 1/3 8 hours later, maximum dose is 7g/day)
  * 25 mg/kg days 2-7
  * 12.5 mg/kg days 8-10
  Interventions: Drug: Ribavirin iv
- Oral favipiravir (Experimental): Oral favipiravir
  * Day 1 2400mg(H0)-2400mg(H8)-1200mg(H16)
  * Day 2-10 1200mg twice daily (BD)
  Interventions: Drug: Favipiravir

INTERVENTIONS:
Drug: Ribavirin iv — 100 mg/kg Day 1 (dose is divided: 2/3 stat, 1/3 8 hours later, maximum dose is 7g/day), then 25 mg/kg days 2-7, 12.5 mg/kg days 8-10
  Other Names: Irrua regimen
  Arms: Intravenous ribavirin
Drug: Favipiravir — Day 1 2400mg(H0)-2400mg(H8)-1200mg(H16), Day 2-10 1200mg twice daily
  Other Names: Avigan
  Arms: Oral favipiravir

SUMMARY:
This exploratory, prospective, controlled, multisite, open label, randomized clinical trial with two treatment arms aims to compare favipiravir, a new treatment candidate for Lassa fever (LF), with the current standard of care, ribavirin.

The primary endpoints of this research are (1) the description of classical pharmacokinetic parameters of favipiravir in comparison with ribavirin standard treatment in patients suffering from LF and (2) the safety and tolerability of both study drugs in the investigated regimens.

DETAILED DESCRIPTION:
The currently used antiviral for the treatment of LF, which is also recommended by the World Health Organization (WHO) and the Nigeria Center for Disease Control, is ribavirin. However, evidence for ribavirin efficacy in LF patients adds up to the results of a single study with serious limitations. A promising new treatment candidate that showed efficacy against LF in preclinical studies is Favipiravir. It has further been evaluated for the treatment of Ebola Virus disease during the West-African Ebola outbreak and is approved for treatment of pandemic influenza virus infections in Japan.

The study will be conducted at two study sites in Nigeria: the Irrua Specialist Teaching Hospital (ISTH) and the Federal Medical Center of Owo (FMCO). Lassa fever patients of 18 years and older with LF confirmed by reverse-transcription polymerase chain reaction (RT-PCR) hospitalized at either ISTH or FMCO will be asked to participate in this study. A total of 40 evaluable participants will be randomized to two treatment arms (20 participants per arm): intravenous ribavirin standard of care treatment (Irrua regimen), oral favipiravir. Patients will be included in the study after giving written informed consent and if all inclusion criteria and no exclusion criteria are met. Multiple blood draws with the purpose of virologic, serologic and immunological analyses, hematological and biochemical analyses as well as pharmacokinetic analyses will be performed throughout the study duration of ten days. Adverse events (AEs), serious adverse events (SAEs) and pregnancy will be captured, monitored and followed-up. A medical monitor will be available for study investigators to assist with any clinical and safety related questions. An external data safety monitoring board (DSMB) will conduct periodic safety reviews.

Data will be captured on source documents and electronic case report forms (eCRFs). Informed consent forms will be stored in a lockable cabinet. Participants data will only be linked to the unique identifier to ensure pseudonymity.

Statistical analysis of study endpoints and pharmacokinetic parameters will be performed descriptively. Missing data will be treated as such, no imputation will be applied.

The study will be conducted in compliance with the protocol, the Declaration of Helsinki, the International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) guideline and the Nigerian National Code for Health Research Ethics, in particular concerning the submission to the ethics committees and the protection of personal data as well as other national and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* LF confirmed by RT-PCR (reverse-transcription polymerase chain reaction)
* Written informed consent

Exclusion Criteria:

* Inability to give consent (e.g. unconscious patients/ cognitively impaired patients)
* Pregnancy/lactation (evidenced by negative urine pregnancy test in women of child-bearing potential)
* Women who plan to get pregnant within the upcoming 6 months
* Severe malnutrition (BMI<16)
* Known intolerance to ribavirin or favipiravir
* History of hemoglobinopathies (i.e., sickle-cell anaemia or thalassemia major) and/or haemophilia
* Organ failure as evidenced by:

  * Creatinine ≥ 3x upper limit of normal (ULN)
  * Aspartate aminotransferase (AST/GOT) > 150 IU/l
  * Alert, confusion, voice, pain, unresponsive (ACVPU) score = V or P or U (corresponds to Glasgow Coma Scale (GCS) ≤ 12)
  * Severe central nervous system features (e.g. seizures, restlessness, confusion and coma)
  * O2 Saturation < 90%
  * Hematocrit <30 %
  * Severe anaemia requiring blood transfusion
* Inability to take oral drug (e.g. encephalopathy, severe vomiting)
* Patients who already received ribavirin or favipiravir within the preceding 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of favipiravir: Maximum plasma concentration (Cmax) | Day 1, Day 2, Day 4, Day 6, Day 7, Day 8 and Day 10 of the study conduct
  Maximum plasma concentration (Cmax) of favipiravir
Pharmacokinetic parameter of favipiravir: Time to maximum concentration (Tmax) | Day 1, Day 2, Day 4, Day 6, Day 7, Day 8 and Day 10 of the study conduct
  Time to maximum concentration (Tmax) of favipiravir
Pharmacokinetic parameter of favipiravir: Area under the concentration-time curve (AUC) | Day 1, Day 2, Day 4, Day 6, Day 7, Day 8 and Day 10 of the study conduct
  Area under the concentration-time curve (AUC) of favipiravir
Pharmacokinetic parameter of favipiravir: Half life (T1/2) | Day 1, Day 2, Day 4, Day 6, Day 7, Day 8 and Day 10 of the study conduct
  Half life (T1/2) of favipiravir
Proportion of drug related AEs and SAEs of both study treatments | throughout study completion (10 days per participant)
  Safety and tolerability of ribavirin and favipiravir in investigated regimens by investigating the proportion of drug related AEs and SAEs

SECONDARY OUTCOMES:
Mutagenicity | 10 days
  Mutagenicity of ribavirin and favipiravir measured via nucleotide exchange rate in individual Lassa virus genomes
Change from baseline in Viral RNA loads | Day of enrollment - Day 10
  Description of viral loads during treatment Relative Lassa virus RNA concentrations in RNA copies per milliliters (RNA copies/ml).
Change from baseline in Lassa virus titers | Day of enrollment - Day 10
  Description of infectious titers during treatment. Infectious titers expressed as focus forming units per milliliters or FFU/ml using immuno-focus assay for Lassa virus.
Change from baseline in Lassa virus serological status | 10 days
  Description of antibody response during treatment. To evaluate the presence or absence of Lassa virus immunoglobulin M (IgM) and G (IgG) antibodies; qualitative results
Pharmacokinetic (PK) modelling and simulations | Day 1, Day 2, Day 4, Day 6, Day 7, Day 8 and Day 10 of the study conduct
  Dosing regimen (mg/frequency/day) resulting in optimal PK/PD target attainment
Correlation between drug exposure and different parameters | 10 days
  Correlation between drug exposure (AUC, Cl/F) and i. Viral elimination dynamics (elimination rate constant), including time to viral clearance (time to negative RT-PCR blood for Lassa virus), regression analysis of viral loads in function of time ii. Length of hospital stay: duration of hospitalization as defined by the enrollment date to discharged data iii. Number of deaths: mortality records iv. Blood component therapy use as concomittant medication
Co-variates impacting on drug exposure | 10 days
  Co-variates impacting on drug exposure: demographices, biological, clinical and virologic data captured in patient case files and sources documents may be assessed as convariates on drug exposure

CONTACTS AND LOCATIONS:
Overall Officials: Peter Akhideno, Dr, Principal Investigator — ISTH; Sylvanus Okogbenin, Prof, Principal Investigator — ISTH; Oluwafemi Ayodeji, Dr, Principal Investigator — FMCO
Locations (2):
- Nigeria (2):
  - Irrua Specialist Teaching Hospital, Irrua, Edo
  - Federal Medical Center of Owo, Owo, Ondo State

IPD SHARING:
Plan to Share IPD: Yes
In line with the funding conditions, individual participant data (IPD) is to be shared. However, this will be de-identified IPD that used to generate the results reported (text, tables, figures and appendices). IPD sharing will begin after publication of primary results and will be available for a period which is aligned with the data sharing agreements approved by the research ethics committees of the counties/sites participating in the trial. The IPD shall be made available via a request and evaluation process to investigators whose proposed research has received IRB approval. All investigators to whom this IPD is made available will be required to be part of the execution of a data use agreement.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: From the time of publication and for a period which is aligned with the data sharing agreements approved by the research ethics committees of the counties/sites participating in the trial.
Access Criteria: This IPD shall be made available via a request and evaluation process to investigators whose proposed research has received inistitutional review board (IRB) approval. All investigators to whom this IPD is made available will be required to be part of the execution of a data use agreement. The data shall be made available through a governed data access process which includes a transparent, accountability and decision-making process: Completion of data request form Evaluation by a data access committee Data sharing Agreement Secure transfer of data

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT04907682/Prot_ICF_000.pdf